CLINICAL TRIAL: NCT06436365
Title: Is the Expert Nail With Poller Screws Superior to the Distal Tibial Locked Plate in the Management of Short Oblique Distal Tibial Fractures?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Dr., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-190-2020
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Tibia Fracture
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Intervention Model Description: The authors performed a prospective randomized controlled trial by including 42 patients to compare expert IMN with poller screws (Group One including 21 patients) versus distal tibial locked plate (Group Two including 21 patients) in fixation of extra-articular distal tibial fractures. The study was conducted after obtaining clearance from the Scientific Board and the Ethical Committee and all patients signed informed consents before starting the study.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- expert IMN with poller screws (Experimental): Twenty-one patients underwent IMN fixation by placing in a supine position with the knee flexed at 90 degrees above the radiolucent table to enable intraoperative imaging and a bolster was put below the thigh to enable knee flexion up to 110 degrees. Multiple interlocking screws were inserted in the expert nail which costed the double compared to the ordinary nail.
  Interventions: Procedure: Locking expert intramedullary nail fixation
- distal tibial locked plate (Active Comparator): patients underwent distal locked plates by placing in a supine position and raising of the contralateral iliac crest which enhanced the rotation and made it easier for medial side access. Thigh was elevated and torniquet was put up to 300 mmHg. By reduction preservation, proximal screws were inserted by small incisions which was followed by insertion of the remained distal screws.
  Interventions: Procedure: Distal locked plate

INTERVENTIONS:
Procedure: Locking expert intramedullary nail fixation — the fracture was reduced to enable the insertion of the guide wire to restore the rotation, length, and angulation. Poller screws were used as control deformity by narrowing the medullary canal and were inserted on the deformity concave side between the nail and bone cortex. A ball-ended guidewire was placed through the entry point to the tibial canal and then to the tibial fracture site under the guidance of fluoroscopy. The guide wire should be inserted centrally within the distal segment on both lateral and anteroposterior views and be far about 1 to 0.5 centimeters from the ankle joint. Reamers with deep fluted and small diameters were used slowly to increase the diameter to reach 0.5 mm till the cortical chatter.
  The nail was inserted by attachment of insertion device and locking of the proximal screw to the nail by directing its apex posteriorly. The nail insertion was done by flexing the knee to prevent any patellar impingement.
  Arms: expert IMN with poller screws
Procedure: Distal locked plate — Cobb dissector was used in creation extra-periosteal subcutaneous tunnel for gentle introduction of a proper plate which was determined by choosing appropriate size and level guided by imaging which helped in prevention of any periosteal damage. Manual closed reduction was performed using the percutaneous clamps. Distal screws were positioned as the following, one was inserted above the medial malleolus, another one was inserted right and below the fracture, and the other screws were inserted to help in anatomical plate positioning. By reduction preservation, proximal screws were inserted by small incisions which was followed by insertion of the remained distal screws.
  Arms: distal tibial locked plate

SUMMARY:
Distal tibial fracture management is difficult because of poor blood supply resulted from subcutaneous location. Therefore, the study aims to compare expert intramedullary nail (IMN) with poller screws to the distal tibial locked plate regarding operative and complications outcomes

DETAILED DESCRIPTION:
Stabilization of the fractured segments is the main goal in fracture fixation which will help to achieve proper healing, fasten early mobility, and get the full function of the injured limb. The fractures may be managed conservatively or by fixation whether internal or external .

Tibial fractures are the most common long bone fractures because of their subcutaneous location which makes them more liable to trauma. They are more common in young males as they are related to sports and traffic accidents. Elderly people come in second place of tibial fractures because they are more likely to occur from simple falls. Proper surgical management of displaced tibial fracture will help in increasing bone stability with the surrounding tissue and improving the bone alignment which in turn fastens the early movement, increases overall function, and prevents prolonged bedridden.

Distal tibia fractures represent from 7% to 10% of all lower limb fractures. Basically, there is controversy over the use of the term "distal tibial fractures" Some authors use the term to describe the distal metaphyseal fractures as defined by one Muller square as Giannoudis 2015 et al. Others use distal tibial fractures to refer to distal shaft fractures (meta-diaphyseal region) from 4 to 11 centimeters starting from the plafond as Polat 2015 et al . Others use the term for both regions, describing them as " two muller squares" as Mauffrey 2012 et al.

Management of distal tibial fracture management is difficult especially in old patients with mature skeletons and without involvement of knee joint because of a fracture near the position to the ankle joint with decreased blood flow resulting from the subcutaneous anatomical location [8]. There are common fixation techniques performed in distal tibial fracture management like open reduction with internal fixation, intramedullary nail insertion (IMN), minimally invasive percutaneous plate osteosynthesis, and external fixation with limited open reduction and internal fixation.

Despite these different management methods achieving success in proper reduction and enhancing the stability and union, they were associated with disadvantages that need to be considered during the management plan which makes no single method ideally preferred for all combined bone and soft tissue distal tibial traumas. Therefore, studies should address all advantages, disadvantages, and the proper application of each method.

We aim in our study to compare expert IMN with poller screws to the distal tibial locked plates in the management of the short oblique distal tibial fractures regarding clinical outcomes, radiological findings, complications, and the need for a secondary operation.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature (18-60 years) male and female patients presented with short oblique fractures which were defined by a fracture with an oblique fracture line its an inclination equal to or greater than 30° with respect to the perpendicular to the axis of the tibia .

Exclusion Criteria:

* We excluded patients presented with other fracture patterns
* intraarticular distal tibial fractures, old fractures, infected fractures, open fractures, and pathological fractures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Olerud Molander Ankle Score (OMAS) | 2 weeks
  questionnaire assessing main nine aspects (daily life activity, pain, supports, swelling, jumping, stiffness, squatting, stair climbing, and running) with a maximum score of 100 indicated normal and minimal score of zero indicated totally impaired function. The score was graded by excellent (for scores between 91 to 100), good (scores between 61 to 90), fair (scores between 31 to 60), and poor (scores between 0 to 30)

SECONDARY OUTCOMES:
Complications | 2 weeks and 6 months
  Complications were also assessed like malunion, delayed union, deep venous thrombosis, infection, and nonunion.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital - Faculty of Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No